CLINICAL TRIAL: NCT02532660
Title: Fase III Study to Evaluate the Efficacy of LABCAT TCJUSS in Patients With Depressive Episode
Brief Title: Study to Evaluate the Efficacy of LABCAT TCJUSS in Patients With Depressive Episode
Acronym: LABCATTCJUSS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Recruitment difficulties due to monocentric study
Sponsor: Laboratório Catarinense SA (Industry)
Collaborators: Universidade Federal do Ceara (Other); Financiadora de Estudos e Projetos (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Laboratório Catarinense Ltda
Record Dates: First submitted 2015-08-23; First posted 2015-08-26 (Estimated); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Escitalopram + LABCAT TCJUSS (Experimental): Escitalopram 10mg + LABCAT TCJUSS 1000 mg daily (two 250mg capsules in the morning + 2 capsules of 250 mg at night);
  Interventions: Drug: Escitalopram 10mg; Drug: LABCAT TCJUSS
- Escitalopram + LABCAT TCJUSS placebo (Placebo Comparator): Escitalopram 10mg + LABCAT TCJUSS placebo daily (2 capsules in the morning + 2 capsules at night);
  Interventions: Drug: Escitalopram 10mg; Drug: LABCAT TCJUSS Placebo
- Escitalopram Placebo + LABCAT TCJUSS (Experimental): Escitalopram Placebo + LABCAT TCJUSS 1000 mg daily (2 capsules in the morning + 2 capsules at night).
  Interventions: Drug: LABCAT TCJUSS; Drug: Escitalopram Placebo

INTERVENTIONS:
Drug: Escitalopram 10mg — Escitalopram 10mg (1 pill once a day)
  Arms: Escitalopram + LABCAT TCJUSS; Escitalopram + LABCAT TCJUSS placebo
Drug: LABCAT TCJUSS — LABCAT TCJUSS 1000mg daily (two 250mg capsules in the morning + 2 capsules of 250 mg at night)
  Arms: Escitalopram + LABCAT TCJUSS; Escitalopram Placebo + LABCAT TCJUSS
Drug: LABCAT TCJUSS Placebo — LABCAT TCJUSS placebo daily (2 capsules in the morning + 2 capsules at night);
  Arms: Escitalopram + LABCAT TCJUSS placebo
Drug: Escitalopram Placebo — Escitalopram Placebo (1 pill once a day)
  Arms: Escitalopram Placebo + LABCAT TCJUSS

SUMMARY:
Evaluate the therapeutic effects of Escitalopram versus an association of Escitalopram + Trichilia catigua Dry Extract (LABCAT TCJUSS) in the average alteration on depression score measured by the Hamilton Scale (HAM-D).

DETAILED DESCRIPTION:
Evaluate the therapeutic effects of Escitalopram versus an association of Escitalopram + LABCAT TCJUSS in the following aspects:

1. Alteration on the average score of anhedonia symptoms through the Shaps-C Scale;
2. Alteration of average scores of Global Clinical Impression carried out by the investigator (CGI-S e CGI-I);
3. Average scores of the Patient Global Evaluation

ELIGIBILITY:
Inclusion Criteria:

* Subjects from both sexes aged between 18 and 65 years;
* Patient diagnosed with mild depression episode confirmed by psychiatric and psychometric evaluation, presenting basal scores above 08 and below 24 measured by the Hamilton Rating Scale (HAM-D);
* Capable of understanding the nature and objective of the study, including risks and adverse effects and intended to cooperate with the researcher and act in accordance with the requirements of the entire protocol, which comes to be confirmed by signing the informed consent.

Exclusion Criteria:

* Have a known hypersensitivity to Trichilia catigua or history of serious adverse reactions;
* Shows risk of suicide, assault, murder or moral exposure;
* Clinical history of bleeding disorders;
* Drug addiction, including alcohol;
* Known or suspected neoplasia;
* Knowledge positive test result for the human immunodeficiency virus;
* Patient not willing to adhere to the procedures of the Protocol;
* For women, can not be pregnant or nursing and must be in use of a contraception method during the participation in the study;
* Patients using other drugs with sedative or antidepressant action, which can not be suspended for 15 days (wash out);
* Diabetics;
* Hyperthyroidism;
* Participation in any experimental study or use of any experimental drug three months before the start of this study;
* Has any condition which the investigator deems relevant to the non-participation of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
HAM-D SCORE REDUCTION | WEEKS 2 (Visit 2), 4 (Visit 3), 8 (Visit 4) and 10 (Visit 5)
  A comparison will be performed between groups in mean reduction in the HAM-D score between baseline (V1-D1) and at weeks 2 (V2), 4 (V3), 8 (V4) and 10 (V5) treatment, following the primary and secondary described outcomes.

SECONDARY OUTCOMES:
Evaluation of symptoms of anhedonia by the change in mean score of Shaps-C scale of pleasure | WEEKS 2 (Visit 2), 4 (Visit 3), 8 (Visit 4) and 10 (Visit 5)
Change in mean scores of Clinical Global Impression performed by the investigator (CGI-I - Improvement) | WEEKS 2 (Visit 2), 4 (Visit 3), 8 (Visit 4) and 10 (Visit 5)
Change in mean scores of Clinical Global Impression performed by the investigator (CGI-S - Severity) | WEEKS 2 (Visit 2), 4 (Visit 3), 8 (Visit 4) and 10 (Visit 5)
Change in mean scores of Global Patient Evaluation scale | WEEKS 2 (Visit 2), 4 (Visit 3), 8 (Visit 4) and 10 (Visit 5)
Change in mean scores of the of Arizona Sexual Experiences scale (ASEX) | WEEKS 2 (Visit 2), 4 (Visit 3), 8 (Visit 4) and 10 (Visit 5)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Elisabete Moraes, Principal Investigator — Universidade Federal do Ceara (UFC)
Locations (1):
- Unidade de Farmacologia Clínica (UNIFAC - Universidade Federal do Ceará), Fortaleza, Ceará, Brazil